CLINICAL TRIAL: NCT03823261
Title: Effects of a Nurse-delivered Cognitive Behaviour Therapy on Adherence and Depressive Symptoms in HIV Infected Persons of South Korea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2018-0755
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, open-label cohort study without a control, and no blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — HIV(+) Koreans with depressive symptoms or poor adherence are our target population. This study is a hospital based implementation research. Most PLWH in South Korea regularly visit ID clinics in tertiary hospitals. The ID clinic of study site can reach the target population. In the clinic, the levels of adherence are routinely measured, and depressive symptoms will be asked with key questions We plan to enroll 50 subjects for CBT-AD intervention. In addition, 2 nurses who providing CBT service, and 6 health care workers will be enrolled for survey for providers and healthcare workers.

SUMMARY:
Cognitive behaviour therapy (CBT) has repeatedly been found to effectively treat depression in adult populations, and CBT for adherence and depression (CBT-AD) is an effective treatment for improving depressive symptoms and medication adherence in the context of various chronic health conditions, including HIV-infection. However, the effects of CBT have not been evaluated in South Korea. Even though HIV infection is currently a controllable disease for patients on successful antiretroviral therapy, people living with HIV (PLWH) are still suffering from internal and external stigmatization in many Asian countries, including South Korea. It is not clear whether CBP-AD would be successful intervention among Asian countries with cultural background of strong stigmatization on HIV/AIDS. We plan to do survey on facilitators or barriers to patients and providers to identify significant contextual factors in South Korea. Demographic data and clinical data including CD4+ T cell counts, viral loads, and antiretroviral therapy regimens will be collected, as well.

Specialists such as psychiatrist or clinical psychologist would be the best provider for CBT intervention. However, an effective and feasible therapy model should be integrated into primary HIV care in South Korea. Medical personnel within most HIV clinics in South Korea include infectious diseases doctors, clinical nurses, and counselling nurses, but CBT services from psychiatrist or clinical psychologist are not routinely available in many hospitals. Hospital-based counselling services with experienced nurses have been provided in many HIV clinics in South Korea, and the counselling nurses would be feasible providers for CBT intervention of this study. So, we plan to investigate the effects of a nurse-delivered cognitive behaviour therapy.

ELIGIBILITY:
Inclusion criteria:

1. HIV(+) Koreans, using ART
2. Adult (19+ years)
3. Having self-reported depressive symptoms or self-reported adherence<90%
4. Being fluent in Korean

Exclusion criteria:

1. Suicidal ideation
2. Active psychosis
3. Uncontrolled neurological problem
4. Having been initiated on or had their dose of psychotropic medication altered within the past 3 months
5. Currently receiving psychotherapy for depression
6. Having previously received CBT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Level of depression | 1 year
  Individual patient would be measured by Beck depression inventory.
Level of adherence | 1 year
  Individual patient would be measured by visual analog scale and pill counting.

SECONDARY OUTCOMES:
Quality of life | 1 year
  Individual patient would be measured by PozQoL. PozQoL is a tool measuring quality of life among people with HIV.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Infectious Diseases, Department of Internal Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Kim JM, Ye M, Lee JI, Na S, Lee Y, Short D, Choi JY. Implementation of a Nurse-Delivered Cognitive Behavioral Therapy for Adherence and Depression of People Living with HIV in Korea. Infect Chemother. 2022 Dec;54(4):733-743. doi: 10.3947/ic.2022.0118. Epub 2022 Nov 11. PMID 36450289